CLINICAL TRIAL: NCT06089564
Title: Enhancing Oral Hygiene in Children With Hearing Impairment: The Impact of Skit Video Interventions - A Randomized Controlled Trial
Brief Title: Effectiveness of Skit Video to Improve Oral Hygiene Status of Children With Hearing Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Maria Moin, Assistant Professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DowUHS 1
Record Dates: First submitted 2023-09-19; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Hearing Impaired Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Skit video (Active Comparator): The video was shown to children lasting for 5 minutes. It was about oral habits, good and bad food. Video was also showed brushing technique.
  Interventions: Behavioral: Skit video, Pictorial, Sign language
- Pictorial (Active Comparator): The pictures related to brushing technique and oral health advices such as good and bad habits was provided in the form of laminated cards. The children has taken those cards along with them.
  Interventions: Behavioral: Skit video, Pictorial, Sign language
- Signed Language (No Intervention): The oral health education related to oral habits, good and bad food was delivered via sign language with the help of children sign language teacher.

INTERVENTIONS:
Behavioral: Skit video, Pictorial, Sign language — Three oral health educational intervention groups, group A (skit video), group B (pictorial) and group C (sign language) by using Sequentially Numbered Sealed Opaque Envelopes (SNOSE). Children picked a sealed envelope randomly and assigned to oral health education intervention group A, B and C. Participants in group A were assigned a skit video method of oral hygiene intervention and shown 5 minute video on what to eat and how to brush their teeth. The video included that what is good and bad for teeth, and how to brush which includes method, time and duration of tooth brushing. Participants assigned to group B and C was provided same instructions for tooth brushing and eating habits in the form of pictures and sign language respectively. The children of Group A received instructions in the form of laminated cards and asked to take with them at home. Participants in group C were received instructions in sign language in the presence of teacher.
  Arms: Pictorial; Skit video

SUMMARY:
Introduction: Oral health is considered as a vital component of overall health and its importance in children may not be disregarded. In children with hearing impairment, communication barriers may hamper their understanding of oral hygiene practices, making them particularly vulnerable to dental problems. Objective: The objective of this study was to compare effectiveness of skit video, pictorial and sign language interventions to improve oral hygiene status of children with hearing impairment. Methods: Sixty children were completed the study and allocated randomly into each group with twenty children as follows: group A: Skit video, group B: Pictorial, and group C: Sign language. Mean gingival and OHI scores were recorded before and after implementation of interventions. Oral hygiene habits, oral hygiene and gingival index scores were recorded by structured questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Children with hearing impairment and total hearing loss at birth
* Aged 7 to 20 years for both genders,
* Minimum of 20 teeth in the oral cavity
* Children with mild, moderate, and severe gingivitis

Exclusion Criteria:

* Children with dental plaque covered more than two-thirds of their tooth surface, had a plaque score of >1.0
* Children with fair to poor oral hygiene
* Children who had previously participated in any activity or programme promoting oral health within the previous six months
* Children with mild to moderate hearing loss
* Children taking long-term antibiotics
* Children who had used mouthwash within the previous three months
* Children with any known systemic diseases
* Presence of extensive dental calculus
* Uncooperative children

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-07-23 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Plaque Index | one month
  Decrease in mean dental plaque scores from baseline to after intervention
Gingival Index | one month
  Decrease in mean gingival scores from baseline to after intervention

SECONDARY OUTCOMES:
Oral Hygiene Index | One month
  Decrease in mean OHI scores from baseline to after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Maria Moin, MDS, Principal Investigator — Bahria University Dental College
Locations (2):
- Pakistan (2):
  - ABSA School and college for deaf, Karachi, Sindh
  - Ida Rieu College For Blind And Deaf, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No